

(HFH IRB form rev: 02/2012)

| $\Box$ | Δ | т | F |
|------------------|---------------|---|---|
| $\boldsymbol{L}$ | $\overline{}$ | | _ |

MRN:

NAME:

# APPROVAL PERIOD

Feb 28, 2018 - Feb 27, 2019

PROJECT TITLE:

Sleep to Prevent Evolving Affective Disorders (SPREAD) – Stepped Care

INSTITUTIONAL REVIEW BOARD

Christopher Drake, Ph.D. 39450 W. 12 Mile Road Novi, MI 48377

#### 1. WHY IS THIS RESEARCH BEING DONE?

To make reading this consent form easier, the word "you" refers to you throughout the consent form. You have been asked to take part in a research study because you did not achieve relief of your insomnia through the online version of Cognitive Behavioral Therapy for Insomnia (dCBT-I) in the form of the internet application Sleepio. The purpose of the research study is to determine if face-to-face treatment will be effective for insomnia. This therapy for insomnia involves altering sleep patterns in specific ways to improve your ability to fall asleep and stay asleep throughout the night. There will be approximately 60 people including you in this research study at Henry Ford Health System (HFHS).

This study is sponsored by the Robert Wood Johnson Foundation. This means that the sponsor is compensating HFHS for the costs of carrying out this research.

### 2. WHAT WILL HAPPEN IF I TAKE PART IN THIS RESEARCH STUDY?

There will be two groups in the study. The group you are assigned to will be chosen by chance (like flipping a coin). You will have an equal chance of being assigned to each particular group. The groups are: Face-to-Face Cognitive Behavioral Therapy for Insomnia (fCBT-I) and no treatment control group (wait-list).

Your participation in this study will last a total of 8 weeks.

- 1. <u>Face-to-Face Cognitive Behavioral Therapy for Insomnia:</u> This treatment involves a 30 minute intake meeting and 6 one-one-one instructional sessions (~1 hour each) with a sleep specialist who will help you to use specific behavioral techniques, adjustments of sleep habits and ways of thinking about your sleep to improve your ability to fall asleep and stay asleep throughout the night.
- 2. <u>No additional treatment (Control):</u> In this option you will continue to apply the principles and concepts learned through the original dCBT-I. No additional meetings or sessions are required.



(HFH IRB form rev: 02/2012)

| $\Box$ | Δ | т | F |
|------------------|---------------|---|---|
| $\boldsymbol{L}$ | $\overline{}$ | | _ |

MRN:

NAME:

## APPROVAL PERIOD

Feb 28, 2018 – Feb 27, 2019

INSTITUTIONAL REVIEW BOARD

### PROJECT TITLE:

Sleep to Prevent Evolving Affective Disorders (SPREAD) - Stepped Care

We will measure sleep quantity and quality during the study by having you fill out a digital sleep diary that is to be completed every morning during the study. This diary will tell us about your sleep for the night before. This sleep diary will be emailed to you each morning. We will also be assessing your daytime functioning, mood, and sleepiness with questionnaires at the beginning of the study and at the end of the treatment.

#### 3. WHAT ARE THE RISKS OF THE STUDY?

You should tell the person obtaining your consent about any other research studies you are involved in right now. You may experience some sleepiness in any of the protocols and this will be carefully monitored through surveys conducted during the study period. No person's time in bed will be reduced below 5 hours per night. There may be risks or discomforts that are not known at this time.

#### 4. WHAT ARE THE BENEFITS TO TAKING PART IN THE STUDY?

The benefits of participating in this study may include: improvements in the ability to fall asleep and stay asleep throughout the night. You might not be helped by participating in this study. However, others may be helped by what is learned from this research.

#### 5. WHAT OTHER OPTIONS ARE THERE?

You do not have to participate in this study. Your other choices may include:

- Getting treatment for insomnia without being in a study (e.g., receiving drugs to improve your sleep or working with a behavioral sleep specialist in a clinical setting)
- Taking part in another study

Talk to your doctor about your choices before you decide if you will take part in this study.

#### 6. WHAT ABOUT CONFIDENTIALITY?

By signing this consent form, you agree that we may collect, use and release your personal and health information for the purpose of this research study.

We may collect and use:

Your existing medical records.



(HFH IRB form rev: 02/2012)

|--|

MRN:

NAME:

# APPROVAL PERIOD

Feb 28, 2018 - Feb 27, 2019

PROJECT TITLE:

Sleep to Prevent Evolving Affective Disorders (SPREAD) – Stepped Care

INSTITUTIONAL REVIEW BOARD

- New health information created during this study.
- Health insurance and other billing information.

We may release this information to the following people:

- The Principal Investigator and his/her associates who work on, or oversee the research activities.
- Government officials who oversee research (Food and Drug Administration).
- The research sponsor (Robert Wood Johnson Foundation).
- Your insurance company or others responsible for paying your medical bills.
- Other researchers at other institutions participating in the research.

Once your information has been released according to this consent form, it could be released again and may no longer be protected by federal privacy regulations.

This consent form, test results, medical reports and other information about you from this study may be placed into your medical record. Generally, you are allowed to look at your medical record. During the research study, you will not be allowed to look at your research study information that is not in your medical record.

HFHS or others may publish the results of this study. No names, identifying pictures or other direct identifiers will be used in any public presentation or publication about this study unless you sign a separate consent allowing that use.

This consent to use and release your personal and health information will expire at the end of this research study.

You do not have to sign this consent to release your medical information and may cancel it at any time. If you decide not to sign this consent or cancel your consent, you cannot participate in this study. If you notify us that you wish to stop participating in this study, we may continue to use and release the information that has already been collected. To cancel your consent, send a written and dated notice to the principal investigator at the address listed on the first page of this form.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.



(HFH IRB form rev: 02/2012)

| _ | | _ | _ |
|-----------------------|---------------|----|---|
| ١١ | Λ | | _ |
| $\boldsymbol{\omega}$ | $\overline{}$ | ١ı | ᆫ |

MRN:

NAME:

## APPROVAL PERIOD

Feb 28, 2018 – Feb 27, 2019

INSTITUTIONAL REVIEW BOARD

### PROJECT TITLE:

Sleep to Prevent Evolving Affective Disorders (SPREAD) - Stepped Care

#### 7. WHAT IF I AM INJURED?

There is no federal, state, or other program that will compensate you or pay for your medical care if you are injured as a result of participating in this study. You and/or your medical insurance may have to pay for your medical care if you are injured as a result of participating in this study. You are not giving up any of your legal rights by signing this consent form.

### 8. WHO DO I CALL WITH QUESTIONS ABOUT THE STUDY OR TO REPORT AN INJURY?

Christopher Drake, PhD, or his staff member has explained this research study and has offered to answer any questions. If you have questions about the study procedures, or to report an injury you may contact Dr. Drake at 248-344-6672. Medical treatment is available to you in case of an injury.

If you have questions about your rights as a research subject you may contact the Henry Ford Health System IRB Coordinator at (313) 874-4464. The IRB is a group of people who review the research to protect your rights.

#### 9. DO I HAVE TO PARTICIPATE IN THIS STUDY?

No, your participation in this research study is voluntary. If you decide to participate, you can stop at any time. If this happens, you may be asked to return for a visit for safety reasons. You will get the same medical care from HFHS whether or not you participate in this study. There will be no penalties or loss of benefits to which you would otherwise be entitled if you choose not to participate or if you choose to stop your participation once you have started. You will be told about any significant information that is discovered that could reasonably affect your willingness to continue being in the study.

### 10. WHO ELSE CAN STOP MY PARTICIPATION?

The Principal Investigator, sponsor or your doctor can end your participation in the research study at any time. If this happens, you may be asked to return for a visit for safety reasons.



(HFH IRB form rev: 02/2012)

| DATE: |
|-------|
| MRN: |
| NAME: |

# APPROVAL PERIOD

Feb 28, 2018 - Feb 27, 2019

**PROJECT TITLE:** 

Sleep to Prevent Evolving Affective Disorders (SPREAD) – Stepped Care

INSTITUTIONAL REVIEW BOARD

#### 11. WILL IT COST ANYTHING TO PARTICIPATE?

We do not expect there to be any additional costs to you if you participate in this study. Items related to the <u>routine</u> medical care that you would receive even if you did not participate in this study will be billed to you or your insurance company. You have the right to ask what it will cost you to take part in this study.

### 12. WILL I BE PAID TO PARTICIPATE?

If you complete the study, you will be paid a total of \$200. You will be paid by check after the follow-up survey. It takes 3-4 weeks to receive your check after a staff member requests each payment. If you do not finish the study, you will be paid for the part that you did complete.

### 13. CONSENT

You have read this consent form or it has been read to you. You understand what you are being asked to do. Your questions have been answered. Any technical terms you did not understand have been explained to you. You agree to be in this study. You will be given a copy of this consent form.

| Signature of Subject | Date | Time |
|----------------------------------------|------|------|
| Print Name of Subject | _ | |
| Witness to Signature | Date | Time |
| Print Name of Person Obtaining Consent | _ | |
| Signature of Person Obtaining Consent | Date | Time |